CLINICAL TRIAL: NCT01596478
Title: Effectiveness of Cognitive-Motivational Behaviour Therapy in Community
Brief Title: Effectiveness of Therapy Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Problem Gambling Institute of Ontario (Other)
Collaborators: Wayne State University (Other); Windsor Regional Hospital (Other)
Responsible Party: Principal Investigator, Assistant Professor, Wayne State University
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSU-#080211M1F
Record Dates: First submitted 2012-04-26; First posted 2012-05-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2012-05

CONDITIONS: Gambling; Pathological Gambling
Keywords: Gambling; Pathological Gambling
MeSH Terms: conditions — Gambling | interventions — Therapeutics; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment As Usual (Active Comparator): The standard treatment usually provided at the clinic.
  Interventions: Behavioral: Treatment as Usual
- Cognitive Motivational Behavior Therapy (Active Comparator): An approach that addresses motivation to change gambling and behavioral patterns related to gambling.
  Interventions: Behavioral: Cognitive Motivational Behavior Therapy
- 12-week wait list (Active Comparator): Participant will start treatment 12 weeks from day of consent.
  Interventions: Behavioral: 12-week wait list

INTERVENTIONS:
Behavioral: Treatment as Usual — Participants will receive Treatment as Usual, on an individual basis, for 60-minutes once per week for 12 weeks.
  Arms: Treatment As Usual
Behavioral: Cognitive Motivational Behavior Therapy — Participants will receive a combined motivational and cognitive-behavioral therapy, on an individual basis, for 60-minutes once per week for 12 weeks.
  Arms: Cognitive Motivational Behavior Therapy
Behavioral: 12-week wait list — Participants will be randomly assigned to start treatment immediately or to go on a 12-week wait list (where they will start treatment 12 weeks from day of consent).
  Arms: 12-week wait list

SUMMARY:
The efficacy of psychosocial treatments for PG, including cognitive-behaviour therapy (CBT) and motivational interviewing (MI) approaches, has been supported in a handful of clinical trials. Indeed, there is more evidence supporting these two approaches than for any other psychosocial treatment for problem gambling. However, while efficacy studies have been conducted, few studies have examined the effectiveness of behavioural treatment in community-based gambling treatment settings. That is to say, the investigators have a good idea of what works in a laboratory setting (i.e., university research settings), but the investigators have no research assessing the transfer of evidence-based treatments for problem gambling to community care. Efficacy studies provide substantially less information about the actual utility of treatments than do effectiveness trials because the way in which treatment is actually provided in the field (with flexibility in terms of time-frame and technique and the tendency to address co-occurring problems) is different from the much more single-focused (on gambling) way it is conducted in laboratory settings. The proposed study is designed to address this significant gap in the research literature. The investigators propose to conduct a treatment effectiveness trial examining a combined cognitive motivational behavior therapy (CMBT) delivered by community-based problem gambling treatment providers, compared with treatment as usual (TAU).

DETAILED DESCRIPTION:
Pilot Study: Eligible participants will undergo a full consent process and a brief interview to assess demographics. Participants' counselors will be asked to audio-record up to 3 therapy sessions which will subsequently be rated for adherence to CMBT procedures.

Main Study: Eligible participants will undergo a full consent process followed by an in-depth interview, with a research assistant. Following an intake assessment, participants will be randomly assigned to one of the three intervention groups. Randomization also will be balanced based on gender to ensure an equitable distribution of men and women in each condition. The research assistant will give the treatment referrals and will introduce the participant to his/her therapist as appropriate.

Treatment will be provided by clinicians at the Windsor Regional Problem Gambling Services.

* Treatment as usual (TAU) - Therapists will be instructed to conduct therapy as they normally would with PGs entering treatment.
* Cognitive motivational behaviour therapy (CMBT) Therapy will consist of 12 60-minute individual counselling sessions. The cognitive-behavioural portion of the intervention is targeted at addressing gambling-related cognitive distortions (e.g., the idea that the gambler can control random events). Motivational interviewing techniques are included to address participant ambivalence about his/her gambling.

Approximately 8 therapists will provide treatment (4 CMBT and 4 TAU, randomly assigned using flip of a coin.) The therapists enrolled in CMBT will be trained for the study. TAU therapists will be offered training in CMBT once study recruitment goals have been met (thus, eventually all therapists will receive training in CMBT). Prior to providing treatment, therapists selected to administer CMBT will receive intensive training in administration of this approach. The therapists will be selected from the professional staff of the Windsor Regional Hospital's Problem Gambling Services.

-Waitlist control condition (WLC) - WLC participants will wait 12-weeks to begin treatment.

At that point, participants will be randomly assigned to receive TAU or CMBT and will proceed through the same study phase (i.e., treatment and follow-up).

Participants will undergo assessments at intake, post-treatment, 6- and 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Main Study: Participants must score at least a 5 on the NODS, and have gambled in the previous two months. Participants must speak English and be able to provide informed consent.
* Pilot Phase: Participants must be patients of the Problem Gambling Services at Windsor Regional Hospital.

Exclusion Criteria:

* Main Study: Acute psychosis, mania or suicidality for which the participant needs immediate treatment, and current enrollment in formal problem gambling treatment (other than the current admission).
* Participants with a co-occurring psychiatric or substance use condition will receive referrals to appropriate ancillary services.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Changes in pathological gambling severity through treatment | changes in gambling severity from baseline at post-treatment
Changes in problem gambling severity through follow-up | Changes in gambling severity from post-treatment through 6-month and 12-month follow-up periods

SECONDARY OUTCOMES:
Examine putative mechanisms of action of "cognitive motivational behavior therapy" relative to "treatment as usual". | Baseline, and changes in gambling mechanisms of action from baseline at post-treatment, 6 and 12 months after beginning treatment
  Assess treatment motivation, coping style, cognitive distortions, psychiatric severity and gambling self-efficacy before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Ledgerwood, PhD, Principal Investigator — Wayne State University
Locations (1):
- Windsor Regional Hospital Problem Gambling Services, Windsor, Ontario, Canada